CLINICAL TRIAL: NCT06628752
Title: Deep Brain Stimulation for the Treatment of Severe Obsessive-compulsive Disorder
Brief Title: Deep Brain Stimulation for Obsessive-compulsive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-2018
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Deep Brain Stimulation; Randomized Controlled Trial
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and the outcome assessor are blinded to whether the participant receives active or sham stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active stimulation (Active Comparator): Deep brain stimulation - active stimulation
  Interventions: Device: Deep brain stimulation
- Sham stimulation (Sham Comparator): Deep brain stimulation - no stimulation
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Stimulation through a device implanted bilaterally into deep brain structures.

SUMMARY:
The goal of this clinical trial is to evaluate the treatment method of deep brain stimulation (DBS) in patients diagnosed with severe and treatment-resistant obsessive-compulsive disorder (OCD). DBS will be administered into the brain area of the bed nucleus of stria terminalis (BNST).

The main research questions are:

* Does active DBS in BNST reduce OCD symptoms (primary outcome)?
* Does active DBS in BNST reduce anxiety or depressive symptoms and improve the level of daily function?

The participants will be randomized to active or sham DBS in the BNST for six months and we will measure the outcomes before DBS surgery, and six months post-surgery. After the randomization phase, the participants will enter an open-label phase and receive continuous DBS in BNST. Yearly follow-ups will be conducted. The outcomes will be measured through interviews using validated psychometric scales.

ELIGIBILITY:
Inclusion Criteria:

* OCD diagnosed according to the criteria in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV).
* The patients should have received at least 16 sessions of cognitive behavioral therapy, tried three different serotonergic antidepressants in adequate doses for three months, and one serotonergic antidepressant in combination with a neuroleptic drug.
* Severe OCD symptoms: YBOCS ≥ 25 points.
* Substantial incapacity because of his/her symptoms.
* Duration of symptoms: 5 years minimum.
* Understand the consequences of participation in the study and give informed written consent.

Exclusion Criteria:

* Not being able to understand the consequences of the treatment.
* Diagnosed with intellectual disability according to DSM-IV.
* Not meeting the requirements for the neurosurgery procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale, Y-BOCS | From enrollment to the end of treatment after 6 months.
  Validated psychometric scale that measures symptoms of OCD.

SECONDARY OUTCOMES:
Hamilton Anxiety Scale, HAS | From enrollment to the end of treatment after 6 months.
  Validated psychometric scale that measures symptoms of anxiety.
Hamilton Depression scale, HAMD | From enrollment to the end of treatment after 6 months.
  Validated psychometric scale that measures symptoms of depression.
Montgomery Asberg Depression Rating Scale, MADRS | From enrollment to the end of treatment after 6 months.
  Validated psychometric scale that measures symptoms of depression.
Global Assessment of Functioning, GAF | From enrollment to the end of treatment after 6 months.
  Scale that measures level of functioning.
Clinical Global Impression rating scale, CGI | From enrollment to the end of treatment after 6 months.
  Scale that measures symptom improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Patric Blomstedt, Professor, Study Chair — Umeå University
Locations (1):
- Umeå University, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No
We will not share IPD until the study is finished and results are published.